CLINICAL TRIAL: NCT01780766
Title: Whole Body MRI Imaging in Multiple Myeloma at 3 Tesla MRI: What is the Added Value of Diffusion Weighted Imaging in Diagnosis and Follow-up
Brief Title: Whole Body MRI Imaging in Multiple Myeloma at 3 Tesla MRI : Added Value of Diffusion Weighted Imaging
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Steven Pans, Medical Doctor Radiologist, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: FIMM; S51079 (Other: Clinical Trial Centre UZ Leuven)
Record Dates: First submitted 2013-01-26; First posted 2013-01-31 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Multiple Myeloma
Keywords: Whole body MRI; Multiple myeloma; Diffusion Weighted MRI; Whole body scan
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Indolent myeloma patient
- Symptomatic Myeloma patient

SUMMARY:
Whole body MRI with diffusion weighted imaging is a useful imaging tool

* staging and diagnosis
* therapy monitoring All patients will be scanned before and during treatment. The findings on diffusion weighted imaging will be correlated to the golden standard (computer tomography and MRI (T1 and STIR)).

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical and laboratory findings, highly suggestive for multiple myeloma.

Exclusion Criteria:

* All patients who are not allowed to be scanned on MRI (Pacemaker, implants ed.)

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinical and laboratory findings, highly suggestive for multiple myeloma. All patients underwent bone marrow biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-09; Primary Completion 2013-03 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Validation | 2 years
  Validation of whole body MRI diffusion-weighted imaging in multiple myeloma at 3 Tesla MRI: correlation of the new MRI imaging technique (diffusion weighted imaging)to standard validated imaging technique (Computer Tomography and Magnetic Resonance Imaging)

SECONDARY OUTCOMES:
Therapy assessment | 4 years
  Whole body MRI with Diffusion weighted imaging is useful for treatment monitoring in multiple myeloma patients during and after therapy.
  Measurement of apparent diffusion coefficient (ADC) and comparison of ADC before, during and after therapy. Correlation of ADC with clinical findings and standard MRI findings.

OTHER OUTCOMES:
outcome | 5 years
  correlation between early treatment response and outcome of the patient by measuring apparent diffusion coefficient

CONTACTS AND LOCATIONS:
Overall Officials: Steven Pans, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

REFERENCES:
- [Background] Bannas P, Hentschel HB, Bley TA, Treszl A, Eulenburg C, Derlin T, Yamamura J, Adam G, Stubig T, Kroger N, Weber C. Diagnostic performance of whole-body MRI for the detection of persistent or relapsing disease in multiple myeloma after stem cell transplantation. Eur Radiol. 2012 Sep;22(9):2007-12. doi: 10.1007/s00330-012-2445-y. Epub 2012 Apr 29. PMID 22544292